CLINICAL TRIAL: NCT07269678
Title: A Comparative Study of Retroclavicular and Classical Coracoid Infraclavicular Brachial Plexus Blocks Using 0.5% Ropivacaine in Patients Undergoing Forearm Surgery.
Brief Title: Comparative Study of Two Infraclavicular Block Approaches in Forearm Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sargodha Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMC-ANS-2025-001
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Procedure Time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retroclavicular approch (Other): Use of 25 ml 0.5% Ropivacaine via Retroclavicular Approach
  Interventions: Procedure: Retroclavicular infraclavicular brachial plexus block
- Classic coracoid approch (Other): Classic Coracoid Infraclavicular Block with 25 ml 0.5% Ropivacaine
  Interventions: Procedure: Classic coracoid infraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Retroclavicular infraclavicular brachial plexus block — The retro clavicular approach to the Infraclavicular brachial plexus block will be performed by placing probe parasagittally just medial to the coracoid process and caudal from the clavicle. The needle insertion point was located in the supraclavicular fossa, just medial to the shoulder at a point sufficiently posterior to the clavicle and medial to the trapezius muscle insertion point on the clavicle. The needle will be inserted immediately above the clavicle in the space between the coracoid process and the clavicle and advanced from cephalad to caudal.
  Arms: Retroclavicular approch
Procedure: Classic coracoid infraclavicular brachial plexus block — The coracoid approach to the Infraclavicular brachial plexus block will be performed by placing the ultrasound probe parasagittally just medial to the coracoid process and caudal from the clavicle. The needle will be inserted cephalad to the ultrasound probe using an in-plane technique and advanced in a caudal direction toward the posterior aspect of the axillary artery, in the vicinity of the posterior cord of the brachial plexus.
  Arms: Classic coracoid approch

SUMMARY:
It is hypothesized that retro clavicular Infraclavicular brachial plexus block is better than classical coracoid Infraclavicular brachial plexus block in patients undergoing forearm surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 18-60 years.
2. Male Patients
3. Elective forearm surgery
4. BMI ≤30kg/m2
5. American Society of Anesthesiologist (ASA) Physical Status ≤III

Exclusion Criteria:

1. History of known allergy or hypersensitivity against study drug.
2. Previous surgery on the same limb

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-22 (Actual); Primary Completion 2025-08-23 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
1 onset of motor block. | Intraoperatively
  Onset of motor block assess using modified bromage scale
  Score Grade of motor blockade(Modified bromage scale) 0 Normal muscle function with full range of movement of elbow, wrist and fingers .
  1 Decreased muscle power so that patient can move fingers and /or wrist only 2. Complete loss of muscle function with no movement in fingers/wrist
Onset of sensory Block | Intraoperatively l
  Onset of sensory block assess using pin prick method Grade of sensory blockade Score
  1. Feeling sharp pinprick (no block) 0
  2. Blunt sensation on pinprick (partial block 1
  3. No sensation on pinprick (complete block) 2
Block adequate for surgery | Intraoperatively
  Block adequate for surgery when there is no need for local infiltration and general anesthesia
Needle Shadow and shaft visibility using 5 point likert scale. | Intraoperatively
  NEEDLE SHADOW VISIBILITY 5-POINT LIKERT SCALE SCORE Needle tip visibility
  1. Very poor
  2. Poor
  3. Fair
  4. Good
  5. Very good
  5-POINT LIKERT SCALE SCORE Needle Shaft visibility
  1. None of the shaft visualized
  2. Only a small segment of the shaft visualized
  3. Less than half of the shaft visualized
  4. Almost all of the shaft visualized
  5. The entire shaft visualized

SECONDARY OUTCOMES:
Rescue anesthesia requirement | Intraoperatively after regional block
  Rescue anesthesia given when block is not adequate for surgery such as local infiltration and general anesthesia
Complication | Intraoperatively
  Vascular puncture and pneumothorax
Procedure Time | Intraoperatively
  Time from insertion of needle to removal of needle

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Faisal Masood teaching Hospital Sargodha, Sargodha, Punjab Province, Pakistan